CLINICAL TRIAL: NCT04963023
Title: Specific Biomarker Identification of Different Subgroups of Chronic Obstructive Pulmonary Disease
Brief Title: Biomarkers of Chronic Obstructive Pulmonary Disease
Acronym: BIOBPCO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0051
Record Dates: First submitted 2021-06-17; First posted 2021-07-15 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: COPD; Asthma-COPD Overlap Syndrome; Asthma
Keywords: COPD; Asthma-COPD Overlap Syndrome; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome; Asthma | interventions — Restraint, Physical; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- frequent exacerbation patients
  Interventions: Other: Physical examinations; Diagnostic Test: blood test
- non frequent exacerbation patients
  Interventions: Other: Physical examinations; Diagnostic Test: blood test
- Asthma-and-COPD overlap syndrome
  Interventions: Other: Physical examinations; Diagnostic Test: blood test
- Asthmatic patients (without COPD)
  Interventions: Other: Physical examinations; Diagnostic Test: blood test

INTERVENTIONS:
Other: Physical examinations — BPCO physical examinations
Diagnostic Test: blood test — blood test in order to study immunologic markers

SUMMARY:
There are few studies about immunological explorations in COPD. Because of the complications of lung biopsies, analyses are generally made on blood samples instead of lung tissue. No study tried to classify COPD vs Asthma vs ACOS. The investigators wondered if there were differences in biomarkers between these groups. The investigators decided to open a pilot-study among COPD patients followed in Amiens-University Hospital. Each patient will be examined and a blood-test will be performed.

ELIGIBILITY:
Inclusion Criteria:

* BPCO patients
* ACOS patients
* asthmatic patient without BPCO

Exclusion Criteria:

* infection
* exacerbation
* immunosuppressive treatment
* immunosuppressive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic obstructive pulmonary disease (COPD) patients, followed in Amiens-University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
identification specific blood immunologic marker for COPD | one hour
  COPD biomarkers are blood immunologic markers

SECONDARY OUTCOMES:
Complete blood count (CBC) Variation between COPD and asthmatic patients | one hour
c-reactive protein concentration variation between COPD and asthmatic patients | one hour
Plasma protein electrophoresis profile Variation between COPD and asthmatic patients | one hour

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No